CLINICAL TRIAL: NCT00127101
Title: A Phase I Clinical Trial of Oral Suberoylanilide Hydroxamic Acid (Vorinostat; Zolinza) in Combination With Bexarotene in Patients With Advanced Cutaneous T-Cell Lymphoma
Brief Title: An Investigational Study of a Histone Deacetylase (HDAC) Inhibitor Plus Targretin in Cutaneous T-Cell Lymphoma Patients (0683-016)(TERMINATED)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was stopped due to low enrollment.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0683-016; MK0683-016; 2005_019
Record Dates: First submitted 2005-08-02; First posted 2005-08-05 (Estimated); Results first posted 2009-08-14 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Vorinostat; Bexarotene

ARMS (6):
- Cohort 1 (Experimental): Vorinostat 200 milligrams daily for 7 days per week + Bexarotene 150 milligrams/meter[2] daily x 7 days per week
  Interventions: Drug: vorinostat; Drug: Comparator: bexarotene
- Cohort 2 (Experimental): Vorinostat 300 milligrams daily for 7 days per week + Bexarotene 150 milligrams/meter[2] daily x 7 days per week
  Interventions: Drug: vorinostat; Drug: Comparator: bexarotene
- Cohort 2a (Experimental): Vorinostat 200 milligrams daily for 7 days per week + Bexarotene 225 milligrams/meter[2] daily x 7 days per week
  Interventions: Drug: vorinostat; Drug: Comparator: bexarotene
- Cohort 2b (Experimental): Vorinostat 200 milligrams daily for 7 days per week + Bexarotene 300 milligrams/meter[2] daily x 7 days per week
  Interventions: Drug: vorinostat; Drug: Comparator: bexarotene
- Cohort 6 (Experimental): Vorinostat 400 milligrams daily for 7 days per week + Bexarotene 150 milligrams daily for 7 days per week
  Interventions: Drug: vorinostat; Drug: Comparator: bexarotene
- Cohort 7 (Experimental): Vorinostat 400 milligrams daily for 7 days per week + Bexarotene daily for 7 days per week [150 milligrams (Cycle 1) 225 milligrams (Cycle 2-6)
  Interventions: Drug: vorinostat; Drug: Comparator: bexarotene

INTERVENTIONS:
Drug: vorinostat — Dose escalation study starting with vorinostat 200 mg q.d. capsules (1 capsule daily) and rising up to vorinostat 400 mg q.d. capsules (1 capsule daily). Up to 6 months of treatment.
  Other Names: Zolinza
Drug: Comparator: bexarotene — Dose escalation with bexarotene 150 mg/m2 capsules rising up to 300 mg/m2 capsules (1 capsule daily). Up to 6 months of treatment.
  Other Names: Targretin

SUMMARY:
This is an investigational study that increases the dosage to determine the safety/tolerability, and efficacy of a histone deacetylase inhibitor in combination with Targretin in patients with cutaneous T-cell lymphoma in patients who have failed at least one prior systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Women or men greater than or equal to 18 years of age
* Advanced cutaneous T-cell lymphoma, stage IB or higher including Sezary Syndrome with progressive, persistent, or recurrent disease
* Failure of at least one systemic therapy, not including Bexarotene (Targretin)
* Eastern Cooperative Oncology Group (ECOG) status less than or equal to 2 (measurement to determine your ability to perform daily activities)

Exclusion Criteria:

* Patient has had investigational treatment in the preceding 30 days
* Active hepatitis B or C, history of HIV
* Prior treatment with any HDAC inhibitor
* Patients must be disease free from prior malignancies for greater than 5 years, except for curatively treated basal cell or squamous cell carcinoma of the skin or carcinoma in-situ of the cervix

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2005-09; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Dummer R, Beyer M, Hymes K, Epping MT, Bernards R, Steinhoff M, Sterry W, Kerl H, Heath K, Ahern JD, Hardwick JS, Garcia-Vargas J, Baumann K, Rizvi S, Frankel SR, Whittaker SJ, Assaf C. Vorinostat combined with bexarotene for treatment of cutaneous T-cell lymphoma: in vitro and phase I clinical evidence supporting augmentation of retinoic acid receptor/retinoid X receptor activation by histone deacetylase inhibition. Leuk Lymphoma. 2012 Aug;53(8):1501-8. doi: 10.3109/10428194.2012.656625. Epub 2012 Feb 13. PMID 22239668

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 7: Vorinostat 400 milligrams daily for 7 days per week + Bexarotene daily for 7 days per week [150 milligrams (Cycle 1) 225 milligrams (Cycle 2-6)]
Period: Base Protocol
Arm/Group | Cohort 1 | Cohort 2 | Cohort 2a | Cohort 2b | Cohort 6 | Cohort 7
Started | 3 | 5 | 3 | 3 | 5 | 4
Completed | 1 | 1 | 1 | 3 | 3 | 3
Not Completed | 2 | 4 | 2 | 0 | 2 | 1
Not completed — Adverse Event | 0 | 2 | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 1 | 0 | 0 | 1
Period: Continuation Phase
Arm/Group | Cohort 1 | Cohort 2 | Cohort 2a | Cohort 2b | Cohort 6 | Cohort 7
Started | 0 | 0 | 1 | 0 (No patients from the 2b Cohort entered into the extension phase) | 3 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 1 | 0 | 3 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 2a | Cohort 2b | Cohort 6 | Cohort 7 | Total
Number analyzed (Participants) | 3 | 5 | 3 | 3 | 5 | 4 | 23
Age, Customized [Number; unit: participants]
  26-35 years of age | 0 | 0 | 1 | 0 | 1 | 0 | 2
  36-45 years of age | 1 | 1 | 0 | 0 | 0 | 0 | 2
  46-55 years of age | 0 | 0 | 1 | 1 | 1 | 1 | 4
  56-65 years of age | 1 | 1 | 1 | 2 | 3 | 1 | 9
  66-75 years of age | 1 | 1 | 0 | 0 | 0 | 2 | 4
  Over 75 years of age | 0 | 2 | 0 | 0 | 0 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 0 | 2 | 2 | 2 | 9
  Male | 1 | 4 | 3 | 1 | 3 | 2 | 14
Race/Ethnicity [Number; unit: participants]
  Turkish | 0 | 0 | 0 | 1 | 0 | 0 | 1
  White | 3 | 5 | 3 | 2 | 5 | 4 | 22

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) as Determined by the Number of Participants With Dose Limiting Toxicities
Description: Number of patients with Dose Limiting Toxicities (DLT). A DLT is an adverse event that determined the treatment dose level was not tolerable for that patient in Cycle 1.
Time Frame: Day 1 to day 28
Population: All Patients treated
Measure: Number; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 2a | Cohort 2b | Cohort 6 | Cohort 7
Number analyzed (Participants) | 3 | 5 | 3 | 3 | 5 | 3
Participants
  DLT | 0 | 2 | 0 | 0 | 0 | 1
  No DLT | 3 | 3 | 3 | 3 | 5 | 2

2. Secondary Outcome: Number of Participants Who Responded to Treatment
Description: Disease burden as assessed by the pre-specified Severity Weighted Assessment Tool (SWAT) measurement. A Response is defined as equal to or greater than 50% improvement in SWAT score.
  SWAT Score is determined by the Lesions classified as patch, plaque, or tumor. The sum of percent of total body surface area (%TBSA) by lesion type is derived and multiplied by a factor of 1 (for patch), 2 (for plaque), or 4 (for tumor). The skin score total is derived by summing the skin score subtotals for patches, plaques and tumors. The skin score total is dimensionless and can range from 0 to 400
Time Frame: Every 28 days for up to 6 Months of Treatment
Population: All patients treated
Measure: Number; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 2a | Cohort 2b | Cohort 6 | Cohort 7
Number analyzed (Participants) | 3 | 5 | 3 | 3 | 5 | 3
Participants
  Response | 0 | 0 | 0 | 1 | 2 | 1
  No Response | 3 | 5 | 3 | 2 | 3 | 2

ADVERSE EVENTS:
Arm/Group | Cohort 1 | Cohort 2 | Cohort 2a | Cohort 2b | Cohort 6 | Cohort 7
Serious Adverse Events (participants affected / at risk) | 2 | 2 | 1 | 0 | 2 | 1
Other Adverse Events (participants affected / at risk) | 3 | 5 | 3 | 3 | 5 | 4
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Cohort 1 | Cohort 2 | Cohort 2a | Cohort 2b | Cohort 6 | Cohort 7
Pyrexia (General disorders) | 0/3 | 0/5 | 1/3 | 0/3 | 0/5 | 0/4
Hypersensitivity (Immune system disorders) | 0/3 | 1/5 | 0/3 | 0/3 | 0/5 | 0/4
Gastroenteritis (Infections and infestations) | 0/3 | 0/5 | 0/3 | 0/3 | 0/5 | 1/4
Lymph Node Abscess (Infections and infestations) | 1/3 | 0/5 | 0/3 | 0/3 | 0/5 | 0/4
Lymphangitis (Infections and infestations) | 1/3 | 0/5 | 0/3 | 0/3 | 0/5 | 0/4
Pneumonia (Infections and infestations) | 0/3 | 1/5 | 0/3 | 0/3 | 0/5 | 0/4
Fall (Injury, poisoning and procedural complications) | 0/3 | 0/5 | 0/3 | 0/3 | 1/5 | 0/4
Mycosis Fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3 | 0/5 | 0/3 | 0/3 | 1/5 | 0/4
T-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3 | 0/5 | 0/3 | 0/3 | 0/5 | 0/4
Skin Necrosis (Skin and subcutaneous tissue disorders) | 0/3 | 0/5 | 1/3 | 0/3 | 0/5 | 0/4
OTHER ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Cohort 1 | Cohort 2 | Cohort 2a | Cohort 2b | Cohort 6 | Cohort 7
Anaemia (Blood and lymphatic system disorders) | 0/3 | 3/5 | 0/3 | 0/3 | 0/5 | 0/4
Anaemia Megaloblastic (Blood and lymphatic system disorders) | 0/3 | 0/5 | 0/3 | 0/3 | 0/5 | 1/4
Eosinophilia (Blood and lymphatic system disorders) | 1/3 | 0/5 | 0/3 | 0/3 | 0/5 | 0/4
Hypochromic Anaemia (Blood and lymphatic system disorders) | 1/3 | 0/5 | 0/3 | 0/3 | 1/5 | 0/4
Leukopenia (Blood and lymphatic system disorders) | 2/3 | 1/5 | 1/3 | 0/3 | 0/5 | 0/4
Lymphopenia (Blood and lymphatic system disorders) | 2/3 | 1/5 | 0/3 | 0/3 | 0/5 | 0/4
Neutropenia (Blood and lymphatic system disorders) | 1/3 | 1/5 | 1/3 | 0/3 | 0/5 | 1/4
Thrombocythaemia (Blood and lymphatic system disorders) | 0/3 | 1/5 | 0/3 | 0/3 | 0/5 | 0/4
Angina Pectoris (Cardiac disorders) | 0/3 | 1/5 | 0/3 | 0/3 | 0/5 | 0/4
Atrial Fibrillation (Cardiac disorders) | 0/3 | 0/5 | 0/3 | 1/3 | 0/5 | 0/4
Atrioventricular Block First Degree (Cardiac disorders) | 0/3 | 0/5 | 0/3 | 1/3 | 0/5 | 0/4
Atrioventricular Block Second Degree (Cardiac disorders) | 0/3 | 0/5 | 0/3 | 1/3 | 0/5 | 0/4
Bradycardia (Cardiac disorders) | 0/3 | 1/5 | 0/3 | 0/3 | 0/5 | 0/4
Deafness (Ear and labyrinth disorders) | 0/3 | 0/5 | 0/3 | 1/3 | 0/5 | 0/4
Tinnitus (Ear and labyrinth disorders) | 0/3 | 0/5 | 0/3 | 0/3 | 1/5 | 0/4
Vertigo (Ear and labyrinth disorders) | 1/3 | 0/5 | 0/3 | 0/3 | 0/5 | 0/4
Hypothyroidism (Endocrine disorders) | 2/3 | 3/5 | 1/3 | 2/3 | 1/5 | 3/4
Dry Eye (Eye disorders) | 0/3 | 0/5 | 0/3 | 0/3 | 1/5 | 0/4
Eyelid Irritation (Eye disorders) | 0/3 | 0/5 | 0/3 | 0/3 | 1/5 | 0/4
Vitreous Opacities (Eye disorders) | 0/3 | 0/5 | 1/3 | 0/3 | 0/5 | 0/4
Abdominal Pain (Gastrointestinal disorders) | 0/3 | 2/5 | 1/3 | 0/3 | 0/5 | 0/4
Abdominal Pain Upper (Gastrointestinal disorders) | 0/3 | 2/5 | 0/3 | 0/3 | 0/5 | 0/4
Constipation (Gastrointestinal disorders) | 0/3 | 0/5 | 0/3 | 0/3 | 0/5 | 1/4
Diarrhoea (Gastrointestinal disorders) | 0/3 | 3/5 | 0/3 | 0/3 | 1/5 | 1/4
Dry Mouth (Gastrointestinal disorders) | 0/3 | 1/5 | 0/3 | 0/3 | 0/5 | 0/4
Flatulence (Gastrointestinal disorders) | 0/3 | 0/5 | 0/3 | 0/3 | 1/5 | 1/4
Lip Swelling (Gastrointestinal disorders) | 0/3 | 0/5 | 1/3 | 0/3 | 0/5 | 0/4
Nausea (Gastrointestinal disorders) | 0/3 | 1/5 | 0/3 | 0/3 | 3/5 | 2/4
Steatorrhoea (Gastrointestinal disorders) | 0/3 | 1/5 | 0/3 | 0/3 | 0/5 | 0/4
Vomiting (Gastrointestinal disorders) | 0/3 | 1/5 | 0/3 | 0/3 | 1/5 | 0/4
Adverse Drug Reaction (General disorders) | 0/3 | 0/5 | 0/3 | 0/3 | 0/5 | 1/4
Asthenia (General disorders) | 1/3 | 0/5 | 0/3 | 0/3 | 0/5 | 0/4
Chest Discomfort (General disorders) | 0/3 | 0/5 | 1/3 | 0/3 | 0/5 | 0/4
Chills (General disorders) | 0/3 | 0/5 | 0/3 | 0/3 | 0/5 | 1/4
Fatigue (General disorders) | 0/3 | 2/5 | 0/3 | 0/3 | 5/5 | 1/4
Feeling Cold (General disorders) | 0/3 | 1/5 | 0/3 | 0/3 | 0/5 | 0/4
Feeling Hot (General disorders) | 0/3 | 0/5 | 0/3 | 0/3 | 1/5 | 0/4
General Physical Health Deterioration (General disorders) | 0/3 | 0/5 | 0/3 | 0/3 | 1/5 | 0/4
Pain (General disorders) | 0/3 | 2/5 | 0/3 | 1/3 | 0/5 | 0/4
Peripheral Coldness (General disorders) | 0/3 | 1/5 | 0/3 | 0/3 | 0/5 | 0/4
Pyrexia (General disorders) | 0/3 | 1/5 | 0/3 | 0/3 | 0/5 | 0/4
Ulcer (General disorders) | 0/3 | 1/5 | 0/3 | 0/3 | 0/5 | 0/4
Abscess Limb (Infections and infestations) | 1/3 | 0/5 | 0/3 | 0/3 | 0/5 | 0/4
Anogenital Warts (Infections and infestations) | 0/3 | 0/5 | 1/3 | 0/3 | 0/5 | 0/4
Conjunctivitis Infective (Infections and infestations) | 0/3 | 0/5 | 0/3 | 1/3 | 0/5 | 0/4
Gingival Infection (Infections and infestations) | 0/3 | 0/5 | 0/3 | 0/3 | 1/5 | 0/4
Influenza (Infections and infestations) | 1/3 | 0/5 | 0/3 | 0/3 | 0/5 | 0/4
Lymph Gland Infection (Infections and infestations) | 1/3 | 0/5 | 0/3 | 0/3 | 0/5 | 0/4
Nasopharyngitis (Infections and infestations) | 0/3 | 1/5 | 1/3 | 0/3 | 0/5 | 1/4
Oral Herpes (Infections and infestations) | 0/3 | 0/5 | 0/3 | 0/3 | 0/5 | 1/4
Otitis Externa (Infections and infestations) | 0/3 | 0/5 | 0/3 | 0/3 | 1/5 | 0/4
Puncture Site Infection (Infections and infestations) | 0/3 | 0/5 | 0/3 | 0/3 | 1/5 | 1/4
Skin Infection (Infections and infestations) | 0/3 | 0/5 | 0/3 | 0/3 | 1/5 | 0/4
Staphylococcal Skin Infection (Infections and infestations) | 0/3 | 0/5 | 0/3 | 0/3 | 1/5 | 0/4
Superinfection (Infections and infestations) | 0/3 | 1/5 | 0/3 | 0/3 | 2/5 | 0/4
Tooth Infection (Infections and infestations) | 0/3 | 0/5 | 0/3 | 0/3 | 1/5 | 0/4
Urinary Tract Infection Bacterial (Infections and infestations) | 1/3 | 0/5 | 0/3 | 0/3 | 0/5 | 0/4
Blood Cholesterol Increased (Investigations) | 0/3 | 0/5 | 0/3 | 0/3 | 0/5 | 1/4
Blood Creatine Phosphokinase Increased (Investigations) | 0/3 | 0/5 | 0/3 | 0/3 | 0/5 | 1/4
Blood Creatinine Increased (Investigations) | 0/3 | 3/5 | 0/3 | 0/3 | 1/5 | 1/4
Blood Potassium Increased (Investigations) | 0/3 | 0/5 | 0/3 | 0/3 | 1/5 | 0/4
Blood Sodium Increased (Investigations) | 0/3 | 0/5 | 0/3 | 0/3 | 1/5 | 0/4
Blood Triglycerides Increased (Investigations) | 0/3 | 0/5 | 1/3 | 1/3 | 0/5 | 1/4
Blood Urea Increased (Investigations) | 0/3 | 1/5 | 0/3 | 0/3 | 0/5 | 0/4
Body Temperature Increased (Investigations) | 0/3 | 1/5 | 0/3 | 0/3 | 0/5 | 0/4
Electrocardiogram QT Prolonged (Investigations) | 0/3 | 1/5 | 0/3 | 0/3 | 0/5 | 0/4
Electrocardiogram ST Segment (Investigations) | 0/3 | 0/5 | 0/3 | 1/3 | 0/5 | 0/4
Electrocardiogram T Wave Inversion (Investigations) | 0/3 | 0/5 | 0/3 | 1/3 | 0/5 | 0/4
High Density Lipoprotein Decreased (Investigations) | 0/3 | 1/5 | 0/3 | 0/3 | 0/5 | 0/4
Thyroxine Free Decreased (Investigations) | 0/3 | 0/5 | 0/3 | 0/3 | 1/5 | 0/4
Tri-Iodothyronine Free Decreased (Investigations) | 0/3 | 0/5 | 0/3 | 0/3 | 0/5 | 1/4
Weight Decreased (Investigations) | 0/3 | 1/5 | 0/3 | 0/3 | 0/5 | 0/4
Anorexia (Metabolism and nutrition disorders) | 0/3 | 1/5 | 0/3 | 0/3 | 1/5 | 0/4
Decreased Appetite (Metabolism and nutrition disorders) | 0/3 | 0/5 | 0/3 | 0/3 | 2/5 | 1/4
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0/3 | 1/5 | 1/3 | 2/3 | 1/5 | 1/4
Hyperkalaemia (Metabolism and nutrition disorders) | 0/3 | 1/5 | 0/3 | 0/3 | 0/5 | 0/4
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3/3 | 3/5 | 2/3 | 1/3 | 1/5 | 2/4
Hypokalaemia (Metabolism and nutrition disorders) | 0/3 | 1/5 | 0/3 | 0/3 | 0/5 | 0/4
Hypophosphataemia (Metabolism and nutrition disorders) | 0/3 | 0/5 | 0/3 | 0/3 | 1/5 | 0/4
Latent Autoimmune Diabetes In Adults (Metabolism and nutrition disorders) | 0/3 | 0/5 | 0/3 | 0/3 | 1/5 | 0/4
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0/3 | 0/5 | 0/3 | 0/3 | 0/5 | 1/4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0/3 | 0/5 | 0/3 | 0/3 | 1/5 | 0/4
Back Pain (Musculoskeletal and connective tissue disorders) | 1/3 | 1/5 | 1/3 | 0/3 | 0/5 | 0/4
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 0/3 | 0/5 | 0/3 | 0/3 | 0/5 | 1/4
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0/3 | 0/5 | 2/3 | 0/3 | 1/5 | 1/4
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1/3 | 0/5 | 0/3 | 0/3 | 0/5 | 0/4
Myalgia (Musculoskeletal and connective tissue disorders) | 0/3 | 1/5 | 1/3 | 0/3 | 0/5 | 0/4
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3 | 1/5 | 0/3 | 0/3 | 2/5 | 0/4
Ageusia (Nervous system disorders) | 0/3 | 1/5 | 0/3 | 0/3 | 0/5 | 0/4
Dizziness (Nervous system disorders) | 0/3 | 1/5 | 0/3 | 0/3 | 0/5 | 2/4
Dysgeusia (Nervous system disorders) | 0/3 | 0/5 | 0/3 | 0/3 | 2/5 | 0/4
Headache (Nervous system disorders) | 0/3 | 1/5 | 1/3 | 1/3 | 2/5 | 0/4
Hypoaesthesia (Nervous system disorders) | 0/3 | 0/5 | 0/3 | 0/3 | 1/5 | 0/4
Hypogeusia (Nervous system disorders) | 0/3 | 0/5 | 0/3 | 0/3 | 0/5 | 1/4
Lethargy (Nervous system disorders) | 0/3 | 0/5 | 0/3 | 1/3 | 0/5 | 0/4
Mental Impairment (Nervous system disorders) | 0/3 | 0/5 | 0/3 | 0/3 | 1/5 | 0/4
Paraesthesia (Nervous system disorders) | 0/3 | 0/5 | 0/3 | 0/3 | 0/5 | 1/4
Peripheral Sensory Neuropathy (Nervous system disorders) | 1/3 | 0/5 | 0/3 | 0/3 | 0/5 | 0/4
Polyneuropathy (Nervous system disorders) | 0/3 | 0/5 | 0/3 | 0/3 | 1/5 | 1/4
Syncope Vasovagal (Nervous system disorders) | 0/3 | 1/5 | 1/3 | 0/3 | 0/5 | 0/4
Anxiety (Psychiatric disorders) | 0/3 | 1/5 | 0/3 | 0/3 | 0/5 | 0/4
Depressed Mood (Psychiatric disorders) | 0/3 | 0/5 | 0/3 | 0/3 | 1/5 | 1/4
Depression (Psychiatric disorders) | 0/3 | 0/5 | 0/3 | 0/3 | 0/5 | 1/4
Insomnia (Psychiatric disorders) | 0/3 | 0/5 | 0/3 | 0/3 | 1/5 | 0/4
Restlessness (Psychiatric disorders) | 0/3 | 0/5 | 0/3 | 0/3 | 1/5 | 0/4
Sleep Disorder (Psychiatric disorders) | 0/3 | 1/5 | 0/3 | 0/3 | 1/5 | 0/4
Haematuria (Renal and urinary disorders) | 1/3 | 0/5 | 0/3 | 0/3 | 0/5 | 0/4
Polyuria (Renal and urinary disorders) | 0/3 | 1/5 | 0/3 | 0/3 | 0/5 | 0/4
Proteinuria (Renal and urinary disorders) | 0/3 | 1/5 | 0/3 | 0/3 | 0/5 | 0/4
Urinary Retention (Renal and urinary disorders) | 0/3 | 1/5 | 0/3 | 0/3 | 0/5 | 0/4
Cough (Respiratory, thoracic and mediastinal disorders) | 0/3 | 1/5 | 0/3 | 1/3 | 0/5 | 0/4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0/3 | 2/5 | 0/3 | 0/3 | 0/5 | 0/4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0/3 | 0/5 | 0/3 | 0/3 | 1/5 | 0/4
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 0/3 | 1/5 | 0/3 | 0/3 | 0/5 | 0/4
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0/3 | 0/5 | 0/3 | 1/3 | 0/5 | 0/4
Alopecia (Skin and subcutaneous tissue disorders) | 0/3 | 1/5 | 0/3 | 1/3 | 3/5 | 1/4
Alopecia Effluvium (Skin and subcutaneous tissue disorders) | 0/3 | 0/5 | 0/3 | 0/3 | 0/5 | 1/4
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0/3 | 1/5 | 0/3 | 0/3 | 0/5 | 0/4
Dry Skin (Skin and subcutaneous tissue disorders) | 0/3 | 1/5 | 0/3 | 0/3 | 1/5 | 0/4
Night Sweats (Skin and subcutaneous tissue disorders) | 1/3 | 0/5 | 0/3 | 0/3 | 0/5 | 0/4
Onychoclasis (Skin and subcutaneous tissue disorders) | 0/3 | 0/5 | 0/3 | 0/3 | 0/5 | 1/4
Pruritus (Skin and subcutaneous tissue disorders) | 0/3 | 1/5 | 0/3 | 0/3 | 3/5 | 0/4
Skin Burning Sensation (Skin and subcutaneous tissue disorders) | 0/3 | 0/5 | 0/3 | 1/3 | 0/5 | 0/4
Skin Fissures (Skin and subcutaneous tissue disorders) | 0/3 | 0/5 | 0/3 | 0/3 | 0/5 | 1/4
Flushing (Vascular disorders) | 0/3 | 0/5 | 0/3 | 0/3 | 0/5 | 1/4
Hypertension (Vascular disorders) | 0/3 | 0/5 | 0/3 | 0/3 | 0/5 | 1/4
Hypotension (Vascular disorders) | 0/3 | 1/5 | 0/3 | 0/3 | 0/5 | 0/4

LIMITATIONS AND CAVEATS:
Study was discontinued due to low enrollment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.